CLINICAL TRIAL: NCT04386356
Title: Airtraq Video Laryngoscope Versus Macintosh Laryngoscope for Endotracheal Intubation by First Year Anaesthesia Trainee in Nepalese Population: A Comparative Study
Brief Title: A Comparative Study of Airtraq Versus Macintosh Laryngoscope for Endotracheal Intubation by First Year Resident
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Sabin Bhandari, Assistant Professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 490/076/077
Record Dates: First submitted 2020-04-25; First posted 2020-05-13 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication
Keywords: Macintosh laryngoscope, Airtraq video laryngoscope

STUDY DESIGN:
Intervention Model Description: First year anaesthesia trainee are those residents in their first year of anaesthesia training and has not had any prior experience using either laryngoscope. They will be given adequate training and instructions before intubation on patients.
  On the day of surgery, the baseline airway variables and the baseline hemodynamic values will be recorded. An investigator not involved in assessing the patient outcome will open the sealed envelope according to the serial number of the patient enrolled into the study.
  Following standard induction technique of preoxygenation with 100% oxygen, injection fentanyl, injection propofol, injection veruronium and mixture of isoflurane and oxygen, tracheal intubation will then be performed by first year anaesthesia trainee using either Airtraq or Macintosh laryngoscope according to the randomization sequence supervised by an experienced anaesthesiologist and data recorded by an independent observer.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An investigator not involved in assessing the patient outcome will open the sealed envelope according to the serial number of the patient enrolled into the study.Tracheal intubation will then be performed by first year anaesthesia trainee using either Airtraq or Macintosh laryngoscope according to the randomization sequence supervised by an experienced anaesthesiologist and data recorded by an independent observer. The data will be analysed by an investigator not involved in administering anaesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Orotracheal intubation with macintosh laryngoscope (No Intervention): Following standard intubation protocol, tracheal intubation will be performed by first year anaesthesia trainee using Macintosh laryngoscope according to the randomization sequence supervised by an experienced anaesthesiologist and data recorded by an independent observer on one group of patients.
  Duration of intubation attempt, failed intubation, optimization maneuvers required to perform tracheal intubation, glottic view according to the Cormack and Lehane grading will be evaluated. Similarly, the maximum fall in oxygen saturation during intubation, HR, SBP and DBP will be documented immediately following intubation and then every 5 minutes till the end of surgery. The occurrence of minor complications (visible trauma to lip or oral mucosa, and presence of blood on laryngoscope blade), and the postoperative sore throat and hoarseness will be evaluated at the end of surgery in the postoperative recovery room.
- Orotracheal intubation with Airtraq Video Laryngoscope (Active Comparator): Following standard intubation protocol, tracheal intubation will be performed by first year anaesthesia trainee using Airtraq video laryngoscope according to the randomization sequence supervised by an experienced anaesthesiologist and data recorded by an independent observer on one group of patients.
  Duration of intubation attempt, failed intubation, optimization maneuvers required to perform tracheal intubation, glottic view according to the Cormack and Lehane grading will be evaluated. Similarly, the maximum fall in oxygen saturation during intubation, HR, SBP and DBP will be documented immediately following intubation and then every 5 minutes till the end of surgery. The occurrence of minor complications (visible trauma to lip or oral mucosa, and presence of blood on laryngoscope blade), and the postoperative sore throat and hoarseness will be evaluated at the end of surgery in the postoperative recovery room.
  Interventions: Device: Orotracheal intubation with either Macintosh laryngoscope versus Airtraq video laryngoscope

INTERVENTIONS:
Device: Orotracheal intubation with either Macintosh laryngoscope versus Airtraq video laryngoscope — Tracheal intubation will be performed by first year anaesthesia trainee using either Macintosh laryngoscope or Airtraq video laryngoscope according to the randomization sequence supervised by an experienced anaesthesiologist and data recorded by an independent observer on one group of patients.
  Arms: Orotracheal intubation with Airtraq Video Laryngoscope

SUMMARY:
This study evaluates the learning and performance of tracheal intubation by first year anaesthesia trainee in Nepalese population using either Airtraq or Macintosh laryngoscopes.

DETAILED DESCRIPTION:
The airway is primarily a conduit for air to reach the lungs. Maintaining a stable, patent airway is a fundamental element of safe perioperative care for all anesthesiologists. Though maintaining airway patency seems conceptually straightforward, a wide variety of clinical circumstances, patients, and tools can make the task of ensuring a stable, open airway under all clinical conditions extremely challenging.

In spite of endotracheal intubation being a lifesaving skill, problems like delayed intubation, misplaced tracheal tube, or airway trauma are frequently encountered, and can cause death or hypoxic brain damage. The magnitude of problems during airway management constitute 17% of anaesthesia closed claims in UK, with difficult intubation being the most common at a rate of 5%.The American Society of Anesthesiologists' Closed Claims Project (ASACCP) reports that though the proportion of claims for respiratory complications decreased from 34% in the 1970s to 15% in the 1990s, the 'big three' (inadequate ventilation, oesophageal intubation, and difficult tracheal intubation) still accounted for >50% of claims leading to death or permanent brain damage.

Direct laryngoscopy (DL) remains the gold standard technique for securing the airway. Successful DL involves the creation of a new (non-anatomic) visual axis, through maximal alignment of the axes of the oral and pharyngeal cavities and displacement of the tongue that requires manipulations of head, neck and larynx and other stressful movements. These manipulations of the airway have numerous adverse implications including significant hemodynamic disturbances, cervical instability, injury to oral and pharyngeal tissues, and dental damage. It is thus, a complicated technical skill with a variable learning curve and requires regular training, experience, and practice to acquire and maintain.

The video laryngoscope (VL) is a recently developed device with a camera and light source on the tip of its blade that provides indirect glottic view. The Airtraq laryngoscope is a recently developed video laryngoscope. It has an anatomically shaped blade which contains two parallel channels, one, the guiding channel, for the insertion of the endotracheal tube (ETT) and the other, the optical channel, containing a series of lenses, prisms, and mirrors that transfer the image from the illuminated tip to a proximal viewfinder, giving a high-quality wide-angle view of the glottis and surrounding structures.

As compared to DL, Airtraq VL requires the application of lesser force to the base of the tongue and is thus less likely to stimulate stress response and induce local tissue injury, produces less cervical movement, and has a faster learning curve relative to DL. It has also been demonstrated to be beneficial in the difficult airway scenario, when compared with the Macintosh laryngoscope, by reducing the number of failed intubations, the duration of intubation attempts and the amount of airway manipulation required, making them suitable for use by medical personnel who intubate infrequently.

The purpose of this study is to evaluate learning and performance of tracheal intubation by first year anaesthesia trainee using either Airtraq VL or Macintosh laryngoscopes.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I and II
2. Age group 16-65 years of either gender
3. Patient requiring orotracheal intubation under general anaesthesia.

Exclusion Criteria:

1. Patient having respiratory tract (oropharynx, larynx) pathology,
2. Patient with predicted difficult airway (such as mouth opening <2 cm),
3. Patient having gastroesophageal reflux disease, hiatus hernia, and pregnancy.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Time required for tracheal intubation. | From the time of randomization and insertion of the blade of the laryngoscope between the dental arches until the endotracheal tube is placed through the vocal cords upto start of surgery, assessed upto 15 minutes
  Duration of intubation attempt will be defined as the time elapsed from insertion of the blade of laryngoscope between the dental arches until the endotracheal tube is placed through the vocal cords and confirmed by chest rise, auscultation, and square wave capnography

SECONDARY OUTCOMES:
Intubation difficulty scale (IDS) score18 for each device. | From the time of randomization and insertion of the blade of the laryngoscope between the dental arches until the endotracheal tube is placed through the vocal cords upto start of surgery, assessed upto 15 minutes
  Number of attempts >1: N1; Each additional attempts add 1 point Number of operators >1: N2; Each additional operators add 1 point Number of alternative techniques: N3; Each techniques add 1 point Cormack Lehane grade: N4; 0 if successful blind intubation; 1 if grade at first attempt is 1 Lifting force required : N5; 0 if normal force required; 1 if increased force required Laryngeal pressure : N6; 0 if not applied; 1 if applied Vocal cord mobility : N7; 0 if abduction 1 if adduction Total IDS : Sum of scores = N1+N2+N3+N4+N5+N6+N7
Rate of successful placement of endotracheal tube. | From the time of randomization and insertion of the blade of the laryngoscope between the dental arches until the endotracheal tube is placed through the vocal cords upto start of surgery, assessed upto 15 minutes
  Successful placement will be confirmed by chest rise, auscultation, and square wave on capnography.
Number of optimization maneuvers required to perform tracheal intubation. | From the time of randomization and insertion of the blade of the laryngoscope between the dental arches until the endotracheal tube is placed through the vocal cords upto start of surgery, assessed upto 15 minutes
  Optimization maneuvers required to perform tracheal intubation will be assessed on a score of 0 to 2:
  0. No maneuvers required.
  1. External laryngeal pressure.
  2. Use of stylet.
Changes in heart rate before and immediately following intubation. | From the randomization and before intubation to immediately following intubation and every 5 minutes till the end of surgery, upto 1 hour
  The blood pressure will be recorded before intubation and assessed again immediately after intubation, and every 5 minutes till the end of the surgery
Incidence of trauma to the airway. | From the time of randomization and insertion of the blade of the laryngoscope between the dental arches until the endotracheal tube is placed through the vocal cords upto start of surgery, assessed upto 15 minutes
  The occurrence of minor complications (visible trauma to lip or oral mucosa, and presence of blood on laryngoscope blade), and the postoperative sore throat and hoarseness will be evaluated at the end of surgery in the postoperative recovery room.
Changes in systolic, diastolic and mean blood pressure before and immediately following intubation | From the randomization and before intubation to immediately following intubation and every 5 minutes till the end of surgery, upto 1 hour
  The blood pressure will be recorded before intubation and assessed again immediately after intubation, and every 5 minutes till the end of the surgery
Changes in oxygen saturation before and immediately following intubation | From the randomization and before intubation to immediately following intubation and every 5 minutes till the end of surgery, upto 1 hour
  The oxygen saturation will be recorded before intubation and assessed again immediately after intubation, and every 5 minutes till the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sabin Bhandari, MD, Principal Investigator — Assistant Professor, Department of Anaesthesiology and Critical Care
Locations (1):
- B P Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenblatt WH, Sukhupragaran W. Airway management. In: Barash PG, Cullen BF, Stoelting RK, Cahalan MK, Stock MC, Ortega R, editors. Clinical Anesthesia. 7th ed. Philadelphia, PA: Wolters Kluwer Health/Lippincott Williams & Wilkins; 2013. p. 774.
- [Background] Berry JM, Harvey S. Laryngoscopic Orotracheal and Nasotracheal Intubation. In: Benumof and Hagberg"s Airway Management; Hagberg CA, Gabel JC, editors, 3rd ed. Philadelphia, PA: Elsevier/Saunders; 2013. p.346-347.
- [Result] Zafirova Z, Tung A. The Difficult Airway: Definitions and Algorithms. In: Glick DB, Cooper RM, Ovassapian A, editors. The difficult airway. New York: Springer; 2013. p.1.
- [Result] Woodall NM, Benger JR, Harper JS, et al. Airway management complications during anaesthesia, in intensive care units and in emergency departments in the UK. Trends in Anaesthesia and Critical Care. 2012; 2(2), 58-64. doi:10.1016/j.tacc.2012.02.005
- [Result] Metzner J, Posner KL, Lam MS, Domino KB. Closed claims' analysis. Best Pract Res Clin Anaesthesiol. 2011 Jun;25(2):263-76. doi: 10.1016/j.bpa.2011.02.007. PMID 21550550
- [Result] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Result] Cook TM, MacDougall-Davis SR. Complications and failure of airway management. Br J Anaesth. 2012 Dec;109 Suppl 1:i68-i85. doi: 10.1093/bja/aes393. PMID 23242753
- [Result] Macintosh RR. A NEW LARYNGOSCOPE. The Lancet. 1943; 241(6233), 205.
- [Result] Miller RA: A new laryngoscope. Anesthesiology. 1941, 2 (3): 310-316. 10.
- [Result] Chemsian R, Bhananker S, Ramaiah R. Videolaryngoscopy. Int J Crit Illn Inj Sci. 2014 Jan;4(1):35-41. doi: 10.4103/2229-5151.128011. PMID 24741496
- [Result] Niforopoulou P, Pantazopoulos I, Demestiha T, Koudouna E, Xanthos T. Video-laryngoscopes in the adult airway management: a topical review of the literature. Acta Anaesthesiol Scand. 2010 Oct;54(9):1050-61. doi: 10.1111/j.1399-6576.2010.02285.x. Epub 2010 Jul 28. PMID 20887406
- [Result] Maharaj CH, Buckley E, Harte BH, Laffey JG. Endotracheal intubation in patients with cervical spine immobilization: a comparison of macintosh and airtraq laryngoscopes. Anesthesiology. 2007 Jul;107(1):53-9. doi: 10.1097/01.anes.0000267529.71756.f0. PMID 17585215
- [Result] Paolini JB, Donati F, Drolet P. Review article: video-laryngoscopy: another tool for difficult intubation or a new paradigm in airway management? Can J Anaesth. 2013 Feb;60(2):184-91. doi: 10.1007/s12630-012-9859-5. Epub 2012 Dec 12. PMID 23233395
- [Result] Nouruzi-Sedeh P, Schumann M, Groeben H. Laryngoscopy via Macintosh blade versus GlideScope: success rate and time for endotracheal intubation in untrained medical personnel. Anesthesiology. 2009 Jan;110(1):32-7. doi: 10.1097/ALN.0b013e318190b6a7. PMID 19104167
- [Result] Kaplan MB, Hagberg CA, Ward DS, Brambrink A, Chhibber AK, Heidegger T, Lozada L, Ovassapian A, Parsons D, Ramsay J, Wilhelm W, Zwissler B, Gerig HJ, Hofstetter C, Karan S, Kreisler N, Pousman RM, Thierbach A, Wrobel M, Berci G. Comparison of direct and video-assisted views of the larynx during routine intubation. J Clin Anesth. 2006 Aug;18(5):357-62. doi: 10.1016/j.jclinane.2006.01.002. PMID 16905081
- [Result] Maharaj CH, Costello JF, Higgins BD, Harte BH, Laffey JG. Learning and performance of tracheal intubation by novice personnel: a comparison of the Airtraq and Macintosh laryngoscope. Anaesthesia. 2006 Jul;61(7):671-7. doi: 10.1111/j.1365-2044.2006.04653.x. PMID 16792613
- [Result] Dhonneur G, Ndoko S, Amathieu R, Housseini LE, Poncelet C, Tual L. Tracheal intubation using the Airtraq in morbid obese patients undergoing emergency cesarean delivery. Anesthesiology. 2007 Mar;106(3):629-30. doi: 10.1097/00000542-200703000-00027. No abstract available. PMID 17325521
- [Result] Nowicki TA, Suozzi JC, Dziedzic M, Kamin R, Donahue S, Robinson K. Comparison of use of the the Airtraq with direct laryngoscopy by paramedics in the simulated airway. Prehosp Emerg Care. 2009 Jan-Mar;13(1):75-80. doi: 10.1080/10903120802471881. PMID 19145529
- [Result] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Result] Maharaj CH, O'Croinin D, Curley G, Harte BH, Laffey JG. A comparison of tracheal intubation using the Airtraq or the Macintosh laryngoscope in routine airway management: A randomised, controlled clinical trial. Anaesthesia. 2006 Nov;61(11):1093-9. doi: 10.1111/j.1365-2044.2006.04819.x. PMID 17042849
- [Result] Ndoko SK, Amathieu R, Tual L, Polliand C, Kamoun W, El Housseini L, Champault G, Dhonneur G. Tracheal intubation of morbidly obese patients: a randomized trial comparing performance of Macintosh and Airtraq laryngoscopes. Br J Anaesth. 2008 Feb;100(2):263-8. doi: 10.1093/bja/aem346. PMID 18211999
- [Result] Malin E, Montblanc Jd, Ynineb Y, Marret E, Bonnet F. Performance of the Airtraq laryngoscope after failed conventional tracheal intubation: a case series. Acta Anaesthesiol Scand. 2009 Aug;53(7):858-63. doi: 10.1111/j.1399-6576.2009.02011.x. Epub 2009 Jun 3. PMID 19496764
- [Result] Turkstra TP, Pelz DM, Jones PM. Cervical spine motion: a fluoroscopic comparison of the AirTraq Laryngoscope versus the Macintosh laryngoscope. Anesthesiology. 2009 Jul;111(1):97-101. doi: 10.1097/ALN.0b013e3181a8649f. PMID 19512871
- [Result] Chalkeidis O, Kotsovolis G, Kalakonas A, Filippidou M, Triantafyllou C, Vaikos D, Koutsioumpas E. A comparison between the Airtraq and Macintosh laryngoscopes for routine airway management by experienced anesthesiologists: a randomized clinical trial. Acta Anaesthesiol Taiwan. 2010 Mar;48(1):15-20. doi: 10.1016/S1875-4597(10)60004-5. PMID 20434108
- [Result] Koh JC, Lee JS, Lee YW, Chang CH. Comparison of the laryngeal view during intubation using Airtraq and Macintosh laryngoscopes in patients with cervical spine immobilization and mouth opening limitation. Korean J Anesthesiol. 2010 Nov;59(5):314-8. doi: 10.4097/kjae.2010.59.5.314. Epub 2010 Nov 25. PMID 21179292
- [Result] Hirabayashi Y, Seo N. Airtraq optical laryngoscope: tracheal intubation by novice laryngoscopists. Emerg Med J. 2009 Feb;26(2):112-3. doi: 10.1136/emj.2008.059659. PMID 19164621
- [Result] Di Marco P, Scattoni L, Spinoglio A, Luzi M, Canneti A, Pietropaoli P, Reale C. Learning curves of the Airtraq and the Macintosh laryngoscopes for tracheal intubation by novice laryngoscopists: a clinical study. Anesth Analg. 2011 Jan;112(1):122-5. doi: 10.1213/ANE.0b013e3182005ef0. Epub 2010 Nov 3. PMID 21048093
- [Result] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827